CLINICAL TRIAL: NCT06107556
Title: Neuromechanical Characterization of Agonist and Antagonist Muscle Activations in the Lower Limbs During Walking After Central Nervous System Injury
Brief Title: Agonist and Antagonist Muscle Activations in the Lower Limbs During Walking After Central Nervous System Injury
Acronym: NEUROGAIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Emilie Hutin, Director, Henri Mondor University Hospital
Other Study IDs: 2023-A02258-37
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Walking, Difficulty; Spasticity/Paresis
MeSH Terms: conditions — Stroke; Mobility Limitation; Muscle Spasticity; Paresis | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gait analysis — 3D gait analysis with electromyographic measurements

SUMMARY:
The retrospective study investigates the part of responsibility of neuromuscular disorders associated with chronic hemiparesis in walking impairment.

DETAILED DESCRIPTION:
After injury to the central nervous system, walking disorders are associated with complex neuromuscular mechanisms that alter the direction and intensity of the descending control, reflex reactions to kinematic changes and the mechanical components of soft tissues. The dissociated analysis of these mechanisms and their interactions during multi-segmental movements and especially during walking is poorly described. However, a quantified assessment of the responsibility of each of the neuromuscular mechanisms in the functional disorder would guide the choice of treatments. 3D gait laboratories provide kinematic data from synchronized walking to surface electromyograms as part of additional assessments to assist in the follow-up of patients with chronic hemiparesis. Retrospective analysis of these data would help to better characterize muscular activation disorders and passive resistance to movement during walking in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Person who performed tridimensional gait analysis in laboratory
* Person who had a stroke at least 6 months before the gait analysis

Exclusion Criteria:

* Any other neurological pathology or gait disorders
* Botulinum toxin injection in the last 3 months before the gait analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Person with a history of stroke
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-19 (Estimated); Primary Completion 2023-10-19 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Coefficient of antagonist activation | 1 year
  The coefficient of antagonist activation of gastrocnemius medialis and soleus was calculated from EMG data by the ratio between the root mean square amplitude during antagonist effort and maximal agonist effort for the same muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Hutin, Principal Investigator — Hôpitaux Universitaires Henri Mondor
Locations (1):
- Laboratoire Analyse et Restauration du Mouvement, Créteil, France

IPD SHARING:
Plan to Share IPD: No